CLINICAL TRIAL: NCT00669227
Title: Intracoronary Stem Cell Therapy in Patients With Acute Myocardial Infarction - A Randomized, Double-blind, Placebo Controlled Trial (SCAMI)
Brief Title: Intracoronary Stem Cell Therapy in Patients With Acute Myocardial Infarction (SCAMI)
Acronym: SCAMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCAMI 01-04
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): autologous stem cells, Ficoll preparation, intracoronary administration at the same day of bone marrow cell aspiration
  Interventions: Other: autologous stem cells
- 2 (Placebo Comparator): placebo is visually indistinguishable from verum due to integration of autologous erythrocytes, intracoronary administration the same day of bone marrow aspiration
  Interventions: Other: placebo suspension

INTERVENTIONS:
Other: autologous stem cells — intracoronary administration at the same day of cell aspiration using the stop flow technique
  Arms: 1
Other: placebo suspension — intracoronary administration at the same day as cell aspiration
  Arms: 2

SUMMARY:
Autologous stem cells may improve myocardial regeneration after intracoronary administration in patients with acute myocardial infarction. The primary hypothesis of this prospective, placebo-controlled, double-blind trial is that the increase of ejection fraction determined by magnetic resonance imaging between baseline and 6 months follow-up is superior in active treated patients compared to patients receiving placebo. The study includes an integrated pilot phase of 40 patients for evaluation of left ventricular ejection fraction determined by cardiac magnetic resonance imaging. Based on the data of this analysis the final sample size will be calculated. The primary endpoint is the improvement in left ventricular ejection fraction with an assumed 2.5% higher improvement in the cell treated population compared to the placebo treated group.

DETAILED DESCRIPTION:
There is a 2:1 randomization for bone marrow cell therapy versus placebo therapy. Patients will be stratified according to age, localization of myocardial infarction and left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction with time to revascularization >6 hours from symptom start
* clear target vessel
* large myocardial infarction defined as: proximal vessel occlusion, CK > 1000 U/L, myocardial scar in magnetic resonance imaging > 10% of left ventricular muscle mass
* potential prior thrombolysis
* written informed consent

Exclusion Criteria:

* acute myocardial infarction with revascularization within 6 hours after symptom start
* prior myocardial infarction
* no clear target vessel
* contraindication for magnetic resonance imaging (e.g. pacemaker, ICD)
* severely depressed left ventricular ejection fraction (less than 20% in magnetic resonance imaging)
* prior hematologic disease
* prior chemo therapy
* prior stem cell transplantation
* prior treatment with G-CSF
* known alteration of the bone marrow by alcohol or drugs, e.g. agranulocytosis
* local infection of puncture sites

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
difference in left ventricular ejection fraction measured by magnetic resonance imaging at baseline and 6 months follow-up | 6 months

SECONDARY OUTCOMES:
left ventricular ejection fraction measured by magnetic resonance imaging | 1, 3, 12 months
left ventricular enddiastolic volume measured by magnetic resonance imaging | 1, 3, 6, 12 months
left ventricular endsystolic volume measured by magnetic resonance imaging | 1, 3, 6, 12 months
major adverse cardiac events | 1, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD; FESC, Principal Investigator — University of Ulm
Locations (1):
- University of Ulm, Ulm, Germany

REFERENCES:
- [Background] Wohrle J, Merkle N, Mailander V, Nusser T, Schauwecker P, von Scheidt F, Schwarz K, Bommer M, Wiesneth M, Schrezenmeier H, Hombach V. Results of intracoronary stem cell therapy after acute myocardial infarction. Am J Cardiol. 2010 Mar 15;105(6):804-12. doi: 10.1016/j.amjcard.2009.10.060. PMID 20211323
- [Background] Wohrle J, von Scheidt F, Schauwecker P, Wiesneth M, Markovic S, Schrezenmeier H, Hombach V, Rottbauer W, Bernhardt P. Impact of cell number and microvascular obstruction in patients with bone-marrow derived cell therapy: final results from the randomized, double-blind, placebo controlled intracoronary Stem Cell therapy in patients with Acute Myocardial Infarction (SCAMI) trial. Clin Res Cardiol. 2013 Oct;102(10):765-70. doi: 10.1007/s00392-013-0595-9. Epub 2013 Jul 30. PMID 23896972